CLINICAL TRIAL: NCT00803075
Title: TALENT Endoluminal Stent Graft System for the Treatment of Abdominal Aortic Aneurysms
Brief Title: Endovascular Repair of Abdominal Aortic Aneurysms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-11092007-864; IRB Protocol 78033
Record Dates: First submitted 2007-12-04; First posted 2008-12-05 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Aortic Aneurysm, Abdominal
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

INTERVENTIONS:
Device: Endovascular Repair of Abdominal Aortic Aneurysms Using TALENT AAA Stent Graft System

SUMMARY:
The purpose of this study is to determine if it is safe and effective to use the TALENT AAA Stent Graft System as a treatment for AAAs in patients who are also candidates for conventional surgical aneurysm repair.

ELIGIBILITY:
Inclusion Criteria:1. Patient has one of the following:

* Aneurysm >4 cm in diameter, or an aneurysm that has increased in size by 0.5 cm in the last 6-months
* Aneurysm is 1.5 times larger than the diameter of the normal infrarenal aorta or symptomatic
* Aneurysm is saccular
* Penetrating ulcer 2. Patient's vascular dimensions must be in the range that can be safely treated with the stent graft available to the physician at the time of the procedure.

  3. Patient has endovascular access to the aneurysmal site with the Introducer Sheath or Delivery Catheter of the appropriate ize device chosen for treatment.

  4. Patient has anatomic characteristics suitable for endovascular repair. 5. Patient has an immediate life-threatening disease of the abdominal aorta in which there is a reasonable likelihood that death will occur within a matter of months or in which premature death is likely without early treatment.

  6. Patient is American Society of Anesthesiology (ASA) grade 1 through 4. 7. Patient is able and willing to comply with 3 month, 6 month, 1 year and every year thereafter post treatment follow-up requirements.

  8. Patient or patient's legal representative understands and has signed an Informed Consent.
 Exclusion Criteria:1. Patient is pregnant or nursing. 2. Patient is morbidly obese or has other clinical conditions that severely inhibit X-ray visualization of the aorta.

  3. Patient has connective disease. 4. Patient is hypercoagulable. 5. Patient has active systemic infection. 6. Patient is less than 18 years old. 7. Patient has less than a one-year life expectancy. 8. Patient is unwilling or unable to return for follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2002-02 (Actual); Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Delivery success
Deployment success
Stent graft migration
Aneurysm exclusion
Stent graft patency
Device integrity
Major morbidity and mortality
Vessel perforation
Stent graft occlusion
Collateral vessel occlusion
Aneurysm rupture

SECONDARY OUTCOMES:
Technical success
Patency

CONTACTS AND LOCATIONS:
Overall Officials: Christopher K Zarins MD, Principal Investigator — Stanford University; Jason T. Lee, Sub-Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States